CLINICAL TRIAL: NCT03126981
Title: A Randomized, Crossover Trial to Assess the Effects of Replacing Refined Carbohydrates With Almonds on Insulin Sensitivity in Men and Women With Prediabetes.
Brief Title: Effects of Almonds on Insulin Sensitivity in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MB-1701
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Diet, Fat-Restricted; Sugars

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole, natural almonds (Experimental): 1.5 oz of whole, natural almonds
  Interventions: Other: 1.5 oz of whole, natural almonds
- Low-fat, high refined starches/sugars (Placebo Comparator): Low-fat foods,high in refined starches and added sugars
  Interventions: Other: Low-fat, high refined starches/sugars

INTERVENTIONS:
Other: 1.5 oz of whole, natural almonds — 1.5 oz of whole, natural almonds
  Arms: Whole, natural almonds
Other: Low-fat, high refined starches/sugars — Low-fat foods, high in refined starches and added sugars
  Arms: Low-fat, high refined starches/sugars

SUMMARY:
The goal of this clinical trial is to evaluate the effects of consuming 1.5 oz almonds twice daily on insulin sensitivity and markers of cardiometabolic health in men and women with prediabetes.

DETAILED DESCRIPTION:
This is a randomized, controlled, two-period crossover study that includes two screening visits, and two 6-week test periods, separated by a 4-week washout. Subjects consume twice daily, 1.5 oz whole, natural almonds (Active Condition) or low-fat foods high in refined starches and added sugars, matched for energy content to the almonds (Control Condition). The assigned study products will be dispensed with instructions to consume 2 servings (Active Product) or 3 servings (Control Products) each day, starting on day 1. Subjects will be screened for prediabetes at the first screening visits. An intravenous glucose tolerance test (IVGTT) will be completed at baseline and the end of each treatment period. Fasting blood samples will be collected for lipid profile and high-sensitivity C-reactive protein (hs-CRP) measurements at all visits. Additionally, blood will be drawn for measurement of Apolipoprotein B and A1, lipoprotein particles and subfractions, Interleukin 6 (IL-6) and Uric acid at the beginning and the end of each test period. Assessments of vital signs, body weight, evaluation of inclusion and exclusion criteria, medication/supplement use, and adverse effects will be performed throughout the study. Compliance will be assessed through a daily log record, and return of unopened study product.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 25.0-39.9 kg/m2
2. Prediabetic: fingerstick glycated hemoglobin 5.7-6.4% (inclusive), or fasting fingerstick capillary glucose of 100-125 mg/dL (inclusive), or 2-h post-prandial glucose of 140-199 mg/dL.
3. Fasting LDL-C level <200 mg/dL and fasting TG level <400 mg/dL.
4. Judged to be in general good health on the basis of medical history and screening laboratory tests.

Exclusion Criteria:

1. Atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis: peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound], history of myocardial infarction, angina, a revascularization procedure, or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
2. History or presence of clinically important pulmonary (including uncontrolled asthma), endocrine (including type I or type II diabetes mellitus), chronic inflammatory disease (including irritable bowel disease, lupus, rheumatoid arthritis), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric, or biliary disorders.
3. Known allergy, sensitivity, or intolerance to any ingredients in the study foods.
4. Uncontrolled hypertension.
5. Recent history of cancer, except for non-melanoma skin cancer.
6. Recent change in body weight of ± 4.5 kg (9.9 lbs).
7. Recent use of any medications intended to alter the lipid profile (e.g. bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin (drug form), omega-3-ethyl ester drugs, and/or PCSK9 inhibitors, with the exception of the stable use of statins), weight-loss drugs or programs, systemic corticosteroid drugs, unstable use of any antihypertensive medication; medications known to influence CHO metabolism (e.g. adrenergic receptor blockers, diuretics, and/or hypoglycemic medications).
8. Recent use of food/supplements known to influence lipid metabolism (e.g. omega-3 fatty acid supplements (e.g., flaxseed, fish or algal oils) or fortified foods, sterol/stanol products; dietary supplements (red rice yeast supplements; garlic supplements; soy isoflavone supplements; niacin or its analogues at doses >400 mg/d, and irregular or inconsistent use of Metamucil® or viscous fiber-containing supplements.
9. Recent use of antibiotics.
10. Pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
11. Extreme dietary habits (e.g. very low CHO diet, vegan, etc.).
12. Current or recent history, or strong potential, for drug or alcohol abuse.
13. History of a diagnosed eating disorder. -

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity index (SI) | 43 days for each treatment period.
  SI from a short (50-min) intravenous glucose tolerance test (IVGTT) at baseline(day 0) and end of two treatment periods (day 43 of both treatment periods)

SECONDARY OUTCOMES:
Fasting lipoprotein lipids | Up to 43 days for each treatment period.
  Fasting blood samples will be collected for measurements of lipoprotein lipids including: Total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non HDL-C, TC/HDL-C ratio and triglycerides (TG) at all visits.
Apolipoprotein (Apo) B and A1, Lipoprotein subfractions and particles | 43 days for each treatment period
  Fasting blood samples will be collected for measurements of Apo B1 and A1, and lipoprotein subfractions and particles at baseline (day 0) and end of the two treatment periods (day 43)
high-sensitivity C-reactive protein (hs-CRP) | Up to 43 days
  Fasting blood samples will be collected for measurement of hs-CRP at all visits.
Serum Uric acid | 43 days for each treatment period
  Fasting blood samples will be collected to measure serum Uric acid levels at the beginning and end of each treatment periods.
Interleukin-6 (IL-6) | 43 days for each treatment period
  Fasting blood samples will be collected to measure serum IL-6 levels at baseline (day 0) and the end of the two treatment periods (day 43)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (2):
- United States (2):
  - MB Clinical Research, Boca Raton, Florida
  - Illinois Institute for Food Safety and Health (IFSH) at Illinois Instiute of Technology (IIT), Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palacios OM, Maki KC, Xiao D, Wilcox ML, Dicklin MR, Kramer M, Trivedi R, Burton-Freeman B, Edirisinghe I. Effects of Consuming Almonds on Insulin Sensitivity and Other Cardiometabolic Health Markers in Adults With Prediabetes. J Am Coll Nutr. 2020 Jul;39(5):397-406. doi: 10.1080/07315724.2019.1660929. Epub 2019 Sep 16. PMID 31525129